CLINICAL TRIAL: NCT04269031
Title: A Phase I, First-in-Human, Randomized, Single-blind, Placebo-controlled Study to Assess the Safety, Tolerability and Pharmacokinetics of AZD2373 Following Single Ascending Dose Administrations to Healthy Male Subjects of African Ancestry
Brief Title: A First-in-human Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AZD2373 After Single Dose Administration in Healthy Male Subjects of African Ancestry.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: D6800C00001
Record Dates: First submitted 2020-02-12; First posted 2020-02-13 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Healthy Volunteers
Keywords: First-in-Human; Randomized; Single-blind; Placebo controlled; AZD2373; Single Ascending Dose; Sentinel Dosing

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: This study is single-blind (in which the study center staff remain blinded during the clinical conduct of a given cohort) with regard to treatment (AZD2373 or placebo) at each dose level. Study subjects will be blinded to treatment allocation throughout the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort 1 (Experimental): On Day 1, randomized subjects will receive a subcutaneous (SC) injection of AZD2373 dose 1 (6 subjects) or matching placebo (2 subjects).
  Interventions: Drug: AZD2373 subcutaneous injection; Drug: Placebo
- Cohort 2 (Experimental): On Day 1, randomized subjects will receive a SC injection of AZD2373 dose 2 (6 subjects) or matching placebo (2 subjects).
  Interventions: Drug: AZD2373 subcutaneous injection; Drug: Placebo
- Cohort 3 (Experimental): On Day 1, randomized subjects will receive a SC injection of AZD2373 dose 3 (6 subjects) or matching placebo (2 subjects).
  Interventions: Drug: AZD2373 subcutaneous injection; Drug: Placebo
- Cohort 4 (Experimental): On Day 1, randomized subjects will receive a SC injection of AZD2373 dose 4 (6 subjects) or matching placebo (2 subjects).
  Interventions: Drug: AZD2373 subcutaneous injection; Drug: Placebo
- Cohort 5 (Experimental): On Day 1, randomized subjects will receive a SC injection of AZD2373 dose 5 (6 subjects) or matching placebo (2 subjects).
  Interventions: Drug: AZD2373 subcutaneous injection; Drug: Placebo
- Cohort 6 (Experimental): On Day 1, randomized subjects will receive a SC injection of AZD2373 dose 6 (6 subjects) or matching placebo (2 subjects).
  Interventions: Drug: AZD2373 subcutaneous injection; Drug: Placebo

INTERVENTIONS:
Drug: AZD2373 subcutaneous injection — Randomised subjects will receive a single ascending dose of AZD2373 by SC injection (dose 1, dose 2, dose 3, dose 4, dose 5 and dose 6).
Drug: Placebo — Randomised subjects will receive a single ascending dose of placebo (saline solution) by SC injection.

SUMMARY:
This is a Phase 1 study to assess the the safety, tolerability and pharmacokinetics (PK) of AZD2373, following subcutaneous (SC) administration of single ascending doses (SAD) of AZD2373 in healthy male subjects of African ancestry.

DETAILED DESCRIPTION:
This study will be conducted as a single-centre, randomised, placebo-controlled, single-blind study to assess the effect of AZD2373 following ascending dose sequential group design administrations to healthy male subjects of African ancestry. The study will include 6 single dose cohorts with the option to include 2 additional cohorts based on emerging data from preceding cohorts in the study.

Approximately 48 male subjects aged 18 to 55 years at the time of informed consent (inclusive) will be randomized with the aim to have 8 subjects participate in each cohort. Within each cohort, 6 subjects will receive AZD2373 and 2 subjects will receive placebo.

Sentinel dosing will be applied for each cohort and will be divided into 2 groups:

* Group 1 (sentinel group): 1 active, 1 placebo;
* Group 2 (the rest of the cohort): 5 active, 1 placebo. The safety data of up to 72 hours post-dose in Group 1 will be reviewed by the Principal Investigator (PI) before the subjects in Group 2 are dosed.

The study will comprise:

* A Screening Period of maximum 35 days;
* A Treatment Period during which subjects will be resident at the Clinical Unit from the day before investigational medicinal product (IMP) administration (Day -1) until at least 72 hours after IMP administration; discharged from the Clinical Unit on Day 4;
* Follow-up Visits on 1, 1.5, 2, 3, 4, 5, 6, and 8 weeks (Visits 3 to 10); and
* A Final Follow up Visit 10 weeks after the last IMP dose.

The visit occurring at 5 weeks post dose (Visit 5) is optional. The expected duration for any subject participating in the study is approximately 10 weeks (excluding an up to 28-day Screening Period).

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures.
* Healthy male subjects of West African ancestry aged 18 to 55 years (inclusive, at time of informed consent) with suitable veins for cannulation or repeated venipuncture.
* Have a body mass index (BMI) between 18 and 35 kg/m^2 (inclusive) and weigh at least 50 kg and no more than 120 kg (inclusive).
* Provision of signed, written and dated informed consent for study participation which includes mandatory genotyping (study objective). NOTE: If a subject would decline to participate in the mandatory genotyping component of the study, the subject will not be included in the study.

Exclusion Criteria:

* Subjects with known ancestry outside of West Africa.
* History of any clinically important disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
* History or presence of gastrointestinal, hepatic or renal disease or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs.
* Any clinically important illness, medical/surgical procedure or trauma within 4 weeks prior to administration of IMP on Study Day 1.
* Any laboratory values with the following deviations:

  1. Alanine aminotransferase or aspartate aminotransferase greater than upper limit of normal and clinically significant as determined by the PI.
  2. White blood cell (WBC) count < 3.0 x 10^9/L.
  3. Hemoglobin (Hb) below lower limit normal .
* Any clinically important abnormalities in clinical chemistry, hematology or urinalysis results, other than those described above, as judged by the PI.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male 18-55 years
Enrollment: 30 (Actual)
Dates: Start 2020-02-13 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events and/or abnormal findings in vital signs, and/or clinical laboratory assessments and/or physical examination and/or electrocardiogram (ECG) evaluation and/or telemetry and/or injection site reactions | Screening Visit to final Follow-up Visit (Week 10 post last dose)
  To assess adverse events as a variable of safety and tolerability of subcutaneous (SC) single ascending dose (SAD) administrations of AZD2373

SECONDARY OUTCOMES:
Area under plasma concentration-time curve from time zero extrapolated to infinity (AUC) | Visit 2 to final Follow-up Visit (Week 10 post last dose)
  To characterize the PK of AZD2373 following SC SAD administrations of AZD2373.
Area under the plasma concentration curve from time zero to the time of last quantifiable analyte concentration (AUClast) | Visit 2 to final Follow-up Visit (Week 10 post last dose)
  To characterize the PK of AZD2373 following SC SAD administrations of AZD2373.
Area under the plasma concentration-time curve from time zero to 72 hours after dosing [AUC(0-72)] | Visit 2 to final Follow-up Visit (Week 10 post last dose)
  To characterize the PK of AZD2373 following SC SAD administrations of AZD2373.
Area under the plasma concentration-time curve from time zero to 48 hours after dosing [AUC (0-48)] | Visit 2 to final Follow-up Visit (Week 10 post last dose)
  To characterize the PK of AZD2373 following SC SAD administrations of AZD2373.
Observed maximum plasma concentration (Cmax) | Visit 2 to final Follow-up Visit (Week 10 post last dose)
  To characterize the PK of AZD2373 following SC SAD administrations of AZD2373.
Time to reach peak or maximum observed concentration or response following drug administration (tmax) | Visit 2 to final Follow-up Visit (Week 10 post last dose)
  To characterize the PK of AZD2373 following SC SAD administrations of AZD2373.
Half-life associated with terminal slope (λz) of a semi logarithmic concentration-time curve (t½λz) | Visit 2 to final Follow-up Visit (Week 10 post last dose)
  To characterize the PK of AZD2373 following SC SAD administrations of AZD2373.
Apparent total body clearance of drug from plasma after extravascular administration [CL/F] | Visit 2 to final Follow-up Visit (Week 10 post last dose)
  To characterize the PK of AZD2373 following SC SAD administrations of AZD2373.
Apparent volume of distribution during the terminal phase after extravascular administration (Vz/F) | Visit 2 to final Follow-up Visit (Week 10 post last dose)
  To characterize the PK of AZD2373 following SC SAD administrations of AZD2373.
Mean residence time of the unchanged drug in the systemic circulation (MRT) | Visit 2 to final Follow-up Visit (Week 10 post last dose)
  To characterize the PK of AZD2373 following SC SAD administrations of AZD2373.
Terminal elimination rate constant (λz) | Visit 2 to final Follow-up Visit (Week 10 post last dose)
  To characterize the PK of AZD2373 following SC SAD administrations of AZD2373.
Time of the last quantifiable concentration [tlast Ae(0-last)] | Visit 2 to final Follow-up Visit (Week 10 post last dose)
  To characterize the PK of AZD2373 following SC SAD administrations of AZD2373.
Cumulative fraction (%) of dose excreted unchanged into the urine from time zero to the last measured time point [fe(0-last)] | Visit 2 to final Follow-up Visit (Week 10 post last dose)
  To characterize the PK of AZD2373 following SC SAD administrations of AZD2373.
Amount of analyte excreted into the urine from time t1 to t2 [Ae(t1-t2)] | Visit 2 to final Follow-up Visit (Week 10 post last dose)
  To characterize the PK of AZD2373 following SC SAD administrations of AZD2373.
Fraction of dose excreted unchanged into the urine from time t1 to t2 [fe(t1-t2)] | Visit 2 to final Follow-up Visit (Week 10 post last dose)
  To characterize the PK of AZD2373 following SC SAD administrations of AZD2373.
Renal clearance of drug from plasma, estimated by dividing Ae(0-t) by AUC(0-t) where the 0-t interval is the same for both Ae and AUC (CLR) | Visit 2 to final Follow-up Visit (Week 10 post last dose)
  To characterize the PK of AZD2373 following SC SAD administrations of AZD2373.
Apolipoprotein L1 (APOL1) concentrations and change from baseline | Visit 2 to final Follow-up Visit (Week 10 post last dose)
  To assess the effect of SC SAD administrations of AZD2373 on plasma concentrations of APOL1 protein

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Goldwater, Dr., Principal Investigator — PAREXEL Early Phase Clinical Unit Baltimore
Locations (1):
- Research Site, Brooklyn, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Bruggeman LA, Sedor JR, O'Toole JF. Apolipoprotein L1 and mechanisms of kidney disease susceptibility. Curr Opin Nephrol Hypertens. 2021 May 1;30(3):317-323. doi: 10.1097/MNH.0000000000000704. PMID 33767059